CLINICAL TRIAL: NCT06494956
Title: A Prospective, Single-center, Open Clinical Study to Evaluate the Safety of Implantable Rechargeable Computerized Deep Nerve Stimulation Systems in Patients With Primary Parkinson's Disease
Brief Title: To Evaluate the Safety of DBS in Patients With Primary Parkinson's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jiangsu CED Medtech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CER-A-PG-01
Record Dates: First submitted 2024-06-17; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Parkinson Disease Dementia
MeSH Terms: interventions — Drug Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single unit (Experimental): An implantable computer fills the deep nervous system and turns it on for treatment
  Interventions: Procedure: Implant device

INTERVENTIONS:
Procedure: Implant device — A subcutaneous tunnel was established under general anesthesia, the electrode was connected to the stimulator, and the pulse generator was implanted in the skull.

SUMMARY:
To evaluate the safety of implantable rechargeable computer deep nerve stimulation system produced by Jiangsu Changyida Medical Technology Co., Ltd. for patients with primary Parkinson's disease

DETAILED DESCRIPTION:
To evaluate the safety of implantable rechargeable computer deep nerve stimulation system produced by Jiangsu Changyida Medical Technology Co., Ltd. for patients with primary Parkinson's disease

ELIGIBILITY:
Inclusion Criteria:1. Aged 18-70 years old, patients with primary Parkinson's disease;2. The duration of Parkinson's disease is 5 years or more;3. The stage of Hoehn-Yahr in the "off" (without medication) state is 2 or more stages;4. UPDRS motion score ≥30 in "Off" state;5. Good response to dopamine drugs, acute levodopa experiment UPDRS exercise score improvement rate of more than 30% (experimental drug Medoba 250mg);6. The daily drug shutdown period is at least 6 hours, or there are sports complications such as serious transactions, and repeated adjustments of drugs still cannot be effectively improved;7. MMSE score ≥24 points on the simple intelligent mental state Examination Scale;8. Have the ability of independent external charging operation;9. Patients or their family members can fully understand the treatment and sign informed consent;10. The patient had good compliance and was able to meet the requirements of postoperative follow-up.

Exclusion Criteria:1. Have received surgical treatment for Parkinson's disease other than deep brain stimulation, such as stereotactic destruction, cell transplantation, gamma knife, etc.;2. The "off" state has serious language disorders, dysphagia, balance disorders and other midline symptoms;3. There are contraindications for neurosurgery, such as cerebral infarction, hydrocephalus, cerebral atrophy, ventricle enlargement, cerebrovascular sequelae, heart disease, severe thrombocytopenia and other cardiovascular and cerebrovascular diseases;4. Have other concomitant diseases, have or need to implant a pacemaker, defibrillator, cochlear implant, other neurostimulator, or need to undergo frequent magnetic examinations;5. Patients who are abnormally sensitive to temperature or allergic to heat;6. There are concomitant diseases that seriously affect health, such as tumors, serious abnormalities of liver and kidney function (indicators exceeding three times the normal value).7. Patients with anxiety and depression.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Start time assessment: Calculate the start time (no change) per day based on the Parkinson's disease diary | 7 months
  Subjects fill in diary cards
Subjects fill in a diary card after device implantation | 6 months
  Subjects fill in diary cards
Drug dosage evaluation | 7 months
  Subjects fill in diary cards
Charging performance evaluation | 6 months
  Subjects fill in diary cards